CLINICAL TRIAL: NCT02283359
Title: An Investigator Sponsored Phase 1a/1b Trial of Selinexor in Combination With Irinotecan in Patients With Adenocarcinoma of Stomach and Distal Esophagus
Brief Title: Selinexor in Combination With Irinotecan in Adenocarcinoma of Stomach and Distal Esophagus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator left the institution
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17919
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Distal Esophagus; Esophageal; Gastric; Carcinoma; Adenocarcinoma; Stomach; Gastro-esophageal junction; Recurrent; Metastatic; Unresectable
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Carcinoma; Adenocarcinoma; Recurrence; Neoplasm Metastasis | interventions — selinexor; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selinexor in Combination with Irinotecan (Experimental): The first study drug is called selinexor (KPT-330). This drug is taken by mouth on days 1, 3, 8 and 10 of each cycle. The starting dose of selinexor will be dependent on the cohort in which the patient is enrolled into. Level -1: 25 mg/m^2; Level 1: 40 mg/m^2; Level 2: 50 mg/m^2; Level 3: 65 mg/m^2.
  The second drug is called irinotecan. This drug is given as intravenous (IV) infusion on days 1 and 8 of each cycle. Participants will receive the standard recommended dose: 125 mg/m^2.
  Interventions: Drug: Selinexor; Drug: Irinotecan

INTERVENTIONS:
Drug: Selinexor — Selinexor is a potent slowly reversible covalent Selective Inhibitor of Nuclear Export (SINE) that specifically blocks the karyopherin protein Exportin 1 or XPO1.
  Other Names: KPT-330
Drug: Irinotecan — Irinotecan is a topoisomerase inhibitor and is approved by FDA to treat colorectal cancer. It is administered intravenously.
  Other Names: Camptosar

SUMMARY:
The main purpose of this study is to see whether the combination of selinexor (KPT-330) and irinotecan can help people with esophageal or stomach cancer. Researchers also want to find out if the combination of selinexor (KPT-330) and irinotecan is safe and tolerable.

DETAILED DESCRIPTION:
This is an open label, single group, non-randomized, phase I study with cohort expansion that utilizes the standard 3+3 design for dose. The dose of selinexor will be escalated in combination with the standard doses of irinotecan. The maximum tolerated dose (MTD) for study is defined as the highest dose level at which 1 or less of 6 patients experience a dose limiting toxicity DLT.

Once the MTD is reached and/or the recommended dose for expansion is determined, an additional cohort of 15 patients with advanced gastric or esophageal cancer will be accrued to better define the safety and tolerability of the combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed gastric, gastro-esophageal junction or distal esophageal adenocarcinoma (predominant histology) that is recurrent, metastatic or unresectable
* Must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1
* Must have received at least one line but less than three lines of prior systemic therapies and have either progressed or intolerant to prior therapies. Patients who have received adjuvant/neoadjuvant therapy within last one year will be eligible as well.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Life expectancy of greater than 3 months
* Must have normal organ and marrow function
* Women of child-bearing potential (WOCBP) must agree to use dual methods of contraception and have a negative serum pregnancy test at screening. Male participants must use an effective barrier method of contraception if sexually active with a WOCBP. For both male and female participants, effective methods of contraception must be used throughout the study and for three months following the last dose.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Have had chemotherapy, biologic therapy or radiotherapy within 3 weeks prior to entering the study
* Are receiving any other investigational agents for anti-cancer treatment within 3 weeks of starting study medication
* Symptomatic central nervous system (CNS) metastases
* Progression on irinotecan containing regimen
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan
* Major surgery within 2 weeks before cycle 1 Day 1 (C1D1)
* Unstable cardiovascular function
* Patients who are pregnant or lactating
* Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study.
* Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen)
* Any underlying condition that would significantly interfere with the absorption of an oral medication
* > Grade 2 peripheral neuropathy at baseline
* Serious psychiatric or medical conditions that could interfere with treatment
* Concurrent therapy with approved or investigational anticancer therapeutic other than steroids
* History of gastrointestinal perforation and/or fistulae within 6 months prior to C1D1
* Use of strong CYP3A4 inducers or inhibitors within 2 weeks of starting study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 18 months
  The MTD for study is defined as the highest dose level at which 1 or less of 6 patients experience a dose limiting toxicity (DLT).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 18 months
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression will be evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Objective Response Rate (ORR) | Up to 18 months
  Only those participants who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis). Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Best Overall Response | Up to 18 months
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Response will be evaluated using RECIST guideline V 1.1. Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria.
Overall Survival (OS) | Up to 18 months
  Overall Survival is defined as the time period from start of treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Mahipal, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States